CLINICAL TRIAL: NCT04231526
Title: A Window of Opportunity Study of Pembrolizumab in Colon Cancer
Brief Title: Pembrolizumab in Early Stage Colon Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to accrue
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-1411
Record Dates: First submitted 2019-12-20; First posted 2020-01-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — pembrolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM A - Pembrolizumab + Surgery (Experimental)
  Interventions: Drug: Pembrolizumab; Procedure: Surgery
- ARM B - Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Pembrolizumab — 2 cycles of neoadjuvant pembrolizumab (200mg IV every 21 days)
  Arms: ARM A - Pembrolizumab + Surgery
Procedure: Surgery — Standard of care surgery

SUMMARY:
This study will gather information on the safety and effectiveness of pembrolizumab, an immunotherapy drug. The purpose of this study is to target early stage colon cancer before it has developed resistance to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed colon adenocarcinoma.
2. No prior chemotherapy, targeted therapy, or immunotherapy for colon cancer.
3. Deemed to have surgically resectable disease.
4. Archival tissue block containing colon adenocarcinoma must be confirmed available prior to enrollment. MSI testing should be obtained prior to starting therapy.
5. Be willing and able to provide written informed consent/assent for the trial.
6. Be 18 years of age or older on day of signing informed consent.
7. Have a measurable primary lesion by lower endoscopy or CT-imaging with a diameter of 1 or more centimeters.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Have no histologically confirmed disseminated disease by CT or PET-CT staging.
10. Male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
11. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 90 days after the last dose of study treatment.
12. Demonstrate adequate organ function as defined below. All screening labs should be performed within 14 days of treatment initiation.

    * Adequate Organ Function Laboratory Values

      * Hematological
    * Absolute neutrophil count (ANC) - ≥1500/µL
    * Platelets - ≥100 000/µL
    * Hemoglobin - ≥7.0 g/dL or ≥5.6 mmol/La

      * Renal
    * Creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) - ≤1.5 × ULN OR

      * 30 mL/min for participant with creatinine levels >1.5 × institutional ULN

        * Hepatic
    * Total bilirubin - ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * AST (SGOT) and ALT (SGPT) - ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

      * Coagulation
    * International normalized ratio (INR) OR prothrombin time (PT)/ Activated partial thromboplastin time (aPTT) - ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

      * ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
    * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
    * Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test during screening (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Known hypersensitivity to pembrolizumab or any of its excipients.
6. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of planned start of study therapy.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has complications from colon cancer including but not limited to organ fistulas, bleeding and obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To measure the feasibility of neoadjuvant pembrolizumab in early stage colon cancer | 14 months
  Measured using RECIST 1.1

SECONDARY OUTCOMES:
Measure the tumor response in early stage colon cancer after neoadjuvant pembrolizumab | 14 months
  Measured using RECIST 1.1
Measure the immune response in early stage colon cancer after neoadjuvant pembrolizumab | 14 months
  Measured using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois